CLINICAL TRIAL: NCT03674021
Title: The Use of a Visual Decision Aid for Shared Decision Making Among Patients With Chest Pain
Brief Title: Use of Visual Decision Aid for Shared Decision Making in Chest Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID pandemic and suspension of observation unit
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CPC
Record Dates: First submitted 2018-08-26; First posted 2018-09-17 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2021-08

CONDITIONS: Acute Coronary Syndrome; Chest Pain; Myocardial Infarction; Angina Pectoris
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Myocardial Infarction; Angina Pectoris

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial where subjects are stratified by gender and then randomized 1:1 to the intervention (CPC) or control arm (usual care).
Who Masked: Outcomes Assessor
Masking Description: The patient, attending physicians, and study team will not be blinded. Outcomes will be assessed through tracing electronic records as well as telephone calls for those whose electronic records are unobtainable. The outcome assessors will be blinded and will follow a telephone script for follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Patients in the intervention arm will receive the Chest Pain Choice visual aid prior to discussion with their primary physician regarding disposition.
  Interventions: Other: Chest Pain Choice visual aid
- Control Arm (No Intervention): Patients in the control arm will not receive the Chest Pain Choice visual aid and will receive standard care.

INTERVENTIONS:
Other: Chest Pain Choice visual aid — The Chest Pain Choice (CPC) decision aid is a visual aid that was developed to facilitate shared decision-making between physicians and patients who present to the emergency department with chest pain. The visual aid includes a brief description of what tests have been done thus far to assess the patient's risk of MACE, a graphic representation of the risk as calculated based on the HEART score, as well as the evaluation options available. The visual aid has been modified from its original form for the local context in terms of viable options for further evaluation.
  Arms: Intervention Arm

SUMMARY:
This study aims to evaluate the use of the chest pain choice (CPC) decision aid as a tool to facilitate discussion between the patient and his/her attending physician with regard to subsequent management plans. Patients aged 21 years and above with low-risk chest pain, as determined by the HEART score (HEART score 0-3), will be included. The investigator's hypothesis is that incorporating the Chest Pain Choice visual aid in shared decision making can help to reduce unnecessary admissions for low risk chest pain to the observation ward, as well as increase patient knowledge with regards to their own condition.

DETAILED DESCRIPTION:
Chest pain is a common presenting complaint in the Emergency Department (ED). Cardiac testing in low-risk patients poses unnecessary costs and resource utilisation, which may in part be due to clinicians adopting a very-low-risk threshold for discharge without testing.

The Chest Pain Choice (CPC) decision aid is a visual aid that was developed to facilitate shared decision-making between physicians and patients who present to the emergency department with chest pain, and has shown to be effective in increasing patient knowledge and decreasing the rate of admission to an observation unit for cardiac testing, among patients with chest pain who are at low risk for acute coronary syndromes. Shared decision making with the use of this visual aid has been shown in other centres to be associated with greater patient knowledge, greater patient involvement in decision making and less frequent admissions, with no increase in major adverse cardiac events (MACE) due to the intervention.

The visual aid includes a brief description of what tests have been done thus far to assess the patient's risk of MACE, a graphic representation of the risk as calculated based on the HEART score, as well as the evaluation options available. The visual aid has been modified from its original form for the local context in terms of viable options for further evaluation.

This study aims to assess if using a visual decision aid for shared decision making between physician and patient can safely help to decrease unnecessary admissions to the ED observation unit, as well as its impact on patient knowledge, satisfaction, as well as 30-day and 60-day Major Adverse Cardiac Events (MACE).

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years and above
* Have low risk chest pain as defined by the HEART score (0-3 points)
* Be English-literate
* Have an initial serum troponin that is less than the 99th centile of the normal reference population
* Have an initial electrocardiogram that is not suggestive of cardiac ischaemia

Exclusion Criteria:

* Have a HEART score of 4 or more
* Are not English-literate
* Have an elevated initial serum troponin
* Have an initial electrocardiogram that is suggestive of cardiac ischaemia (ST-segment depression or elevation, new onset left bundle brunch block, T-wave inversions, etc.)
* Have known coronary artery disease
* Have a prior plan for cardiac intervention or admission
* Have barriers to outpatient follow-up
* Are prisoners
* Are pregnant
* Are hearing or visually impaired, or are otherwise unable to use the clinical decision aid
* Do not consent to participation in the study

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Admission to the Emergency Department Observation Unit | Index visit
  Admission to the Emergency Department Observation Unit during index emergency department visit

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) at 30 days | 30 days after index visit
  MACE is defined as all-cause mortality, myocardial infarction or coronary revascularisation.
Major Adverse Cardiac Events at 60 days | 60 days after index visit
  MACE is defined as all-cause mortality, myocardial infarction or coronary revascularisation.
Emergency Department Attendance at 30 days | 30 days after index visit
  Repeat attendance to the emergency department
Emergency Department Attendance at 60 days | 60 days after index visit
  Repeat attendance to the emergency department
Stress treadmill electrogram at 30 days | 30 days after index visit
  The presence of stress treadmill electrocardiogram at 30 days post index visit
Stress treadmill electrogram at 60 days | 60 days after index visit
  The presence of stress treadmill electrocardiogram at 60 days post index visit
Stress myocardial perfusion imaging at 30 days | 30 days after index visit
  The presence of stress myocardial perfusion imaging at 30 days post index visit
Stress myocardial perfusion imaging at 60 days | 60 days after index visit
  The presence of stress myocardial perfusion imaging at 60 days post index visit
Stress echocardiogram at 30 days | 30 days after index visit
  The presence of stress echocardiogram at 30 days post index visit
Stress echocardiogram at 60 days | 60 days after index visit
  The presence of stress echocardiogram at 60 days post index visit
Computed tomography of the coronary arteries (CTCA) at 30 days | 30 days after index visit
  The presence of computed tomography of the coronary arteries (CTCA) at 30 days post index visit
Computed tomography of the coronary arteries (CTCA) at 60 days | 60 days after index visit
  The presence of computed tomography of the coronary arteries (CTCA) at 60 days post index visit

CONTACTS AND LOCATIONS:
Locations (1):
- Mui Teng Chua, Singapore, Central, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hess EP, Knoedler MA, Shah ND, Kline JA, Breslin M, Branda ME, Pencille LJ, Asplin BR, Nestler DM, Sadosty AT, Stiell IG, Ting HH, Montori VM. The chest pain choice decision aid: a randomized trial. Circ Cardiovasc Qual Outcomes. 2012 May;5(3):251-9. doi: 10.1161/CIRCOUTCOMES.111.964791. Epub 2012 Apr 10. PMID 22496116
- [Result] Anderson RT, Montori VM, Shah ND, Ting HH, Pencille LJ, Demers M, Kline JA, Diercks DB, Hollander JE, Torres CA, Schaffer JT, Herrin J, Branda M, Leblanc A, Hess EP. Effectiveness of the Chest Pain Choice decision aid in emergency department patients with low-risk chest pain: study protocol for a multicenter randomized trial. Trials. 2014 May 10;15:166. doi: 10.1186/1745-6215-15-166. PMID 24884807

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT03674021/Prot_SAP_000.pdf